CLINICAL TRIAL: NCT03498014
Title: Comparison of Standard Opioid Prescription Versus Prescription Guided by Pharmacogenetic Analysis in Patients With Non-cancerous Chronic Pain.
Acronym: AlgoPGx
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no started
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIMAO/2017-02/JCB-01
Record Dates: First submitted 2018-03-29; First posted 2018-04-13 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Non-cancerous Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prescription as standard (Active Comparator)
  Interventions: Other: Standard opioid prescription
- Pharmacogenetic-guided prescription (Experimental)
  Interventions: Other: Pharmacogenetic analysis allowing personalized opioid prescription

INTERVENTIONS:
Other: Pharmacogenetic analysis allowing personalized opioid prescription — Genotypic of patient to determine optimal opioid treatment (tramadol, codeine or oxycodone)
  Arms: Pharmacogenetic-guided prescription
Other: Standard opioid prescription — Opioid prescription made without reference to patient genetic profile (tramadol, codeine or oxycodone)
  Arms: Prescription as standard

SUMMARY:
The investigators hypothesize that opioid prescription guided by patient pharmacogenetic profile will diminish opioid-associated undesirable effects by 50% and improve medication compliance.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient will be available for all visits
* Patients suffer from non-cancerous chronic pain according to HAS criteria
* Patient not having taking opioids in previous 2 months
* Patient indicated for prescription of opioids (oxycodone, codeine or tramadol) or patient not responding to first line treatment

Exclusion Criteria:

* The subject is participating in an category I interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding
* The patient is likely to procreate and does not use an effective method of contraception (contraceptive ring, surgical contraception, implant, patch, contraceptive pill, male and female condoms, IUD)
* There is a contra-indication for opioid use
* Patient with an addiction risk (score ≥ 8 on ORT scale).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Compare presence/absence undesirable events associated to opioid between groups from predefined list | Month 1
  Presence/absence of at least one undesirable event of at least grade 3 according to list in Annex 17.5 of the protocol
Compare presence/absence undesirable events associated to opioid between groups from predefined list | Month 2
  Presence/absence of at least one undesirable event of at least grade 3 according to list in Annex 17.5 of the protocol
Compare presence/absence undesirable events associated to opioid between groups from predefined list | Month 3
  Presence/absence of at least one undesirable event of at least grade 3 according to list in Annex 17.5 of the protocol
Compare presence/absence undesirable events associated to opioid between groups | Month 1
  Presence/absence of at least one undesirable event of at least grade 3 according to Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Compare presence/absence undesirable events associated to opioid between groups | Month 2
  Presence/absence of at least one undesirable event of at least grade 3 according to Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Compare presence/absence undesirable events associated to opioid between groups | Month 3
  Presence/absence of at least one undesirable event of at least grade 3 according to Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)

SECONDARY OUTCOMES:
Number of undesirable events associated to opioid between groups | Month 1
  Total number of undesirable event of at least grade 3 according to list in protocol
Number of undesirable events associated to opioid between groups | Month 2
  Total number of undesirable event of at least grade 3 according to list in protocol
Number of undesirable events associated to opioid between groups | Month 3
  Total number of undesirable event of at least grade 3 according to list in protocol
Number of undesirable events associated to opioid between groups | Month 1
  Total number of undesirable event of at least grade 3 according to Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Number of undesirable events associated to opioid between groups | Month 2
  Total number of undesirable event of at least grade 3 according to Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Number of undesirable events associated to opioid between groups | Month 3
  Total number of undesirable event of at least grade 3 according to Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Compare clinical therapeutic efficacy between groups | Month 1
  Patient Global Impression of Change (PGIC) score; value between 1-7
Compare clinical therapeutic efficacy between groups | Month 2
  Patient Global Impression of Change (PGIC) score; value between 1-7
Compare clinical therapeutic efficacy between groups | Month 3
  Patient Global Impression of Change (PGIC) score; value between 1-7
Compare patient-reported pain between groups | Day 0
  Visual analog scare 1-10
Compare patient-reported pain between groups | Week 2
  Visual analog scare 1-10
Compare patient-reported pain between groups | Month 1
  Visual analog scare 1-10
Compare patient-reported pain between groups | Month 2
  Visual analog scare 1-10
Compare patient-reported pain between groups | Month 3
  Visual analog scare 1-10
Compare neuropathic pain between groups | Day 0
  DN4 score (Douleur Neuropathique 4 Questions); score between 0-10
Compare neuropathic pain between groups | Month 1
  DN4 score (Douleur Neuropathique 4 Questions); score between 0-10
Compare neuropathic pain between groups | Month 2
  DN4 score (Douleur Neuropathique 4 Questions); score between 0-10
Compare neuropathic pain between groups | Month 3
  DN4 score (Douleur Neuropathique 4 Questions); score between 0-10
Compare benefit/risk ratio of treatment between groups | Month 1
  Overall Benefit of Analgesics Score (OBAS); score between 0-32
Compare benefit/risk ratio of treatment between groups | Month 2
  Overall Benefit of Analgesics Score (OBAS); score between 0-32
Compare benefit/risk ratio of treatment between groups | Month 3
  Overall Benefit of Analgesics Score (OBAS); score between 0-32
Compare quality of life between patients in each group | Day 0
  Quality of life Short Form 12 (SF-12) questionnaire; score between 0-100
Compare quality of life between patients in each group | Month 3
  Quality of life Short Form 12 (SF-12) questionnaire; score between 0-100
Compare medication compliance between groups | Month 1
  Serum concentration of tramadol, codeine or oxycodone and their metabolites by Liquid chromatography-tandem mass spectrometry (LC-MS-MS)
Compare medication compliance between groups | Month 2
  Serum concentration of tramadol, codeine or oxycodone and their metabolites by Liquid chromatography-tandem mass spectrometry (LC-MS-MS)
Compare medication compliance between groups | Month 3
  Serum concentration of tramadol, codeine or oxycodone and their metabolites by Liquid chromatography-tandem mass spectrometry (LC-MS-MS)
Qualitive comparison of medication compliance between groups | Month 1
  Presence/absence of opioids or metabolites in serum
Qualitive comparison of medication compliance between groups | Month 2
  Presence/absence of opioids or metabolites in serum
Qualitive comparison of medication compliance between groups | Month 3
  Presence/absence of opioids or metabolites in serum
Serum concentration of tramadol, codeine or oxycodone and their metabolites by Liquid chromatography-tandem mass spectrometry (LC-MS-MS) | Day 0
  Opioids Risk Tool (ORT): scores of 0-3 (low risk), 4-7 (moderate risk), or ≥ 8 (high risk)
Compare observed medication misuse between groups | Month 1
  Prescription Opioid Misuse Index (POMI)
Compare observed medication misuse between groups | Month 2
  Prescription Opioid Misuse Index (POMI)
Compare observed medication misuse between groups | Month 3
  Prescription Opioid Misuse Index (POMI)
Correlation between predicted phenotype and observed metabolic ratios | Month 1
  Products/substrate ratio measured by high performance liquid chromatography-high resolution mass spectrometry (HPLC-HRMS)
Correlation between predicted phenotype and observed metabolic ratios | Month 2
  Products/substrate ratio measured by high performance liquid chromatography-high resolution mass spectrometry (HPLC-HRMS)
Correlation between predicted phenotype and observed metabolic ratios | Month 3
  Products/substrate ratio measured by high performance liquid chromatography-high resolution mass spectrometry (HPLC-HRMS)
Metabolic profile of patients | Month 1
  Extensive Metaboliser, Intermediate Metaboliser, Poor Metaboliser or Ultra-rapid Metaboliser according to CYP2D6 phenotype and polymorphism of the glucuronyl transferase gene UGT2B7
Metabolic profile of patients | Month 2
  Extensive Metaboliser, Intermediate Metaboliser, Poor Metaboliser or Ultra-rapid Metaboliser according to CYP2D6 phenotype and polymorphism of the glucuronyl transferase gene UGT2B7
Metabolic profile of patients | Month 3
  Extensive Metaboliser, Intermediate Metaboliser, Poor Metaboliser or Ultra-rapid Metaboliser according to CYP2D6 phenotype and polymorphism of the glucuronyl transferase gene UGT2B7
Correlation between saliva and plasma concentration of opioids | Month 1
  Concentration of tramadol, codeine or oxycodone and their metabolites by Liquid chromatography-tandem mass spectrometry (LC-MS-MS)
Correlation between saliva and plasma concentration of opioids | Month 2
  Concentration of tramadol, codeine or oxycodone and their metabolites by Liquid chromatography-tandem mass spectrometry (LC-MS-MS)
Correlation between saliva and plasma concentration of opioids | Month 3
  Concentration of tramadol, codeine or oxycodone and their metabolites by Liquid chromatography-tandem mass spectrometry (LC-MS-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Boyer, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France